CLINICAL TRIAL: NCT02868450
Title: Chronic Infection With Tropheryma Whipplei: Risk Factors Related to the Host
Acronym: WHIPPLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-10; 2013-A00460-45 (Other: ANSM)
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Whipple Infection
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with HLA-DQB1 06 and/or HLA-DRB 13 (Experimental)
  Interventions: Biological: Blood Sample

INTERVENTIONS:
Biological: Blood Sample

SUMMARY:
In 2012, a previous work showed that T. whipplei is a common bacterium detected in various situations. A large part of the population is therefore exposed to a T. whipplei but there is that some people probably with immunological and genetic factors predisposing which develop a disease. The association teams with experience in HLA-typing will allow us to better identify patients with a risk of chronic complication.

The main aim of this study is to evaluate if the HLA-DRB13 and/or HLA-DQB106 typing in patients are risk factors of chronic infection with T. whipplei (defined by classic Whipple disease and/ or, endocarditis and/or encephalitis).

DETAILED DESCRIPTION:
Since the first isolation of a strain of Tropheryma whipplei (T. whipplei) and the development of molecular tools, the natural history of this bacterium continued to clarify. The currently proposed scheme is as follows: after contamination human oral-oral or fecal, patients will develop acute infections such as bacteremia, gastroenteritis and pneumonia. They can then produce specific antibodies. Likely depending on the host-related factors, three types of evolution appear to be possible: (i) some patients eliminate the bacteria and develop specific antibodies. (ii) some patients are chronic carriers of the bacterium with a strong immune response. (iii) Finally, patients develop subacute or chronic infections, with an insufficient immune response or non-existent answer to T. whipplei.

Subacute or chronic infections include Whipple's disease characterized by histological involvement of the small intestine, as well as localized without digestive impairment, such as endocarditis or encephalitis. Despite appropriate antibiotic therapy, patients with Whipple's disease will present relapse (30-40% of patients), but also of re-infection with different genotypes of T. whipplei.

Here the hypothesis is that HLA-DRB 13 and/or HLA-DQB1 06 alleles are associated with the presence of chronic infections with T. whipplei (defined by classic Whipple disease and / or endocarditis and/or encephalitis)

ELIGIBILITY:
Inclusion Criteria:

* Patient with a positive PCR to T. Whipplei diagnostics.
* Patient aged > or = 18 years old.
* Patient who does not declined to have his medical records reviewed for research.
* Patient with health insurance.

Exclusion Criteria:

* Patient minors (age <18 years)
* Pregnant woman, parturient or breastfeeding
* Adult Patient under guardianship .
* Patient deprived of liberty under court order
* Patient refusing to sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2013-06-07 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with HLA-DQB1 06 among patients with a chronic infection with T. whipplei (defined by classic Whipple disease and / or endocarditis and/or encephalitis) versus asymptomatic patients | 1 day
Proportion of patients with HLA-DRB 13 among patients with a chronic infection with T. whipplei (defined by classic Whipple disease and / or endocarditis and/or encephalitis) versus asymptomatic patients | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Catherine GEINDRE, Study Director — Assistance Publiques Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided